CLINICAL TRIAL: NCT04120480
Title: Clinical and Economic Effectiveness of Pharmacogenomic (PGx) Testing in Patients With Polypharmacy
Brief Title: Effectiveness of PGx Testing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: OneOme, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1448074-3
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Polypharmacy
Keywords: Genomics
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Testing (Experimental): Participants randomized to this arm will be sent a kit to collect a genetic sample from a swab of their mouths. The kit will have instructions on how to collect the genetic sample and how to send it in a postage-paid envelope to the testing laboratory (OneOme). OneOme will process the sample and The study pharmacist will scan the results and enter any related information into the participant's KPCO electronic health record. If any changes to the participant's medication(s) are recommended (for example: a dose decrease or increase, stop taking your current medication and start another), the study pharmacist will contact the participant's KPCO prescriber directly to discuss the recommendations. The prescriber may contact the participant to change the participant's medication(s).
  Interventions: Diagnostic Test: Pharmacogenomic test
- Usual Care (No Intervention): Participants randomized to this arm will NOT be tested. They will receive usual care and the research will not involve study visits or in-person contact.

INTERVENTIONS:
Diagnostic Test: Pharmacogenomic test — The RightMed test is an end-to-end solution which includes sample collection, PGx testing services, data analysis, and clinical interpretation that helps prescribers select treatments based on evidence-driven predictions of patient drug response and tolerance. Genetic components of an individual's drug response are well established and often included on FDA medication labels. The RightMed test has incorporated existing evidence to classify the risk and likelihood of an antidepressant working for different patients. Patient results for each medication can fall into one of three categories: 1) Green - use as directed; 2) Yellow - use with caution; and 3) Red - adjust dose or choose alternative mediation.
  Arms: Testing

SUMMARY:
The purpose of this study is to determine the clinical and economic effectiveness of a pharmacogenomic (PGx) approach to prescribing medications in patients with high-risk polypharmacy in an integrated healthcare delivery system.

Investigators hypothesize that patients who receive the RightMed® PGx test from OneOme, LLC with subsequent counseling of their prescribers by a study pharmacist, as needed, on the appropriateness of their prescribed medications will experience lower one-year follow-up healthcare utilization and expenditures compared to control patients who receive usual care.

DETAILED DESCRIPTION:
The purpose of this study is to determine the clinical and economic effectiveness of a pharmacogenomic (PGx) approach to prescribing medications in patients with high-risk polypharmacy in an integrated healthcare delivery system.

Investigators hypothesize that patients who receive the RightMed® PGx test from OneOme, LLC with subsequent counseling of their prescribers by a study pharmacist, as needed, on the appropriateness of their prescribed medications will experience lower one-year follow-up healthcare utilization and expenditures compared to control patients who receive usual care.

Primary Objectives:

1. Healthcare expenditures: 6- and 12-month changes in total healthcare expenditures from the Kaiser Permanente Colorado (KPCO) perspective
2. Healthcare utilization: 6- and 12-month changes in hospitalizations, emergency room visits, medical office visits, and telephone encounters

Secondary Objectives:

1. Medication changes: Counts of 6-month medication and/or dose adjustments in targeted medications
2. Medication congruence: Description of counts of RightMed test recommendations accepted by prescribers
3. Medication adherence: 6- and 12-month changes in percent of days (PDC) covered for targeted medications
4. Pharmacy expenditures: 6- and 12-month changes in outpatient prescription medication expenditures from the KPCO perspective

ELIGIBILITY:
Inclusion Criteria:

1. 18-79 years of age
2. Days supply of 5+ medications with 2+ advisable for PGx on the RightMed test
3. English or Spanish speaker
4. Current KPCO member
5. Dispensing 1 med (for advisable for PGx) in the 90 days prior with no dispensing in the previous six months -or- daily dose change (up or down) in the 90 days
6. Prescriber from Smoky Hill, Westminster, Hidden Lake, Skyline, East Denver, or Lakewood clinics
7. Available email address -

Exclusion Criteria:

1. Pregnant (HCG+ test in the previous 9 months)
2. A live birth in the previous 24 months
3. SNF or hospice stay in the previous 1 month
4. Hospitalization in previous 14 days
5. Diagnosis of dementia, delerium, alzheimer's, or parkinson's in the previous 6 months
6. On the KPCO No Contact List -

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Healthcare expenditures | 6 and 12 months after consent
  Changes in mean/median total healthcare expenditures from the KPCO perspective
Healthcare utilization | 6 and 12 months after consent
  Changes in the proportion with at least one and mean/median count of hospitalization, emergency room visit, medical office visit, and telephone encounter

SECONDARY OUTCOMES:
Medication changes | 6 months after consent
  Mean/median counts of medication and/or dose adjustments in targeted medications
Medication congruence | 6 months after consent
  Description of counts of RightMed test recommendations accepted by prescribers
Medication adherence | 6 and 12 months after consent
  Mean/median changes in percent of days (PDC) covered for targeted medications
Pharmacy expenditures | 6 and 12 months after consent
  Mean/median changes in outpatient prescription medication expenditures from the KPCO perspective

CONTACTS AND LOCATIONS:
Overall Officials: Alison Quinn, PharmD, Principal Investigator — KPCO
Locations (1):
- Central Support Services, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No